CLINICAL TRIAL: NCT00200356
Title: Edaravone-Sodium Ozagrel (Thromboxane A2 Synthase Inhibitor) Comparative Post-Marketing Study on Acute Ischemic Stroke
Brief Title: Edaravone-Sodium Ozagrel Comparative Post-Marketing Study on Acute Ischemic Stroke
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Tanabe Pharma Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MCI186-13
Record Dates: First submitted 2005-09-12; First posted 2005-09-20 (Estimated); Results first posted 2013-01-15 (Estimated); Last update posted 2026-01-07 (Actual); Status verified 2025-12

CONDITIONS: Cerebral Infarction
MeSH Terms: conditions — Cerebral Infarction | interventions — Edaravone; ozagrel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Edaravone (Experimental)
  Interventions: Drug: Edaravone
- Ozagrel (Active Comparator)
  Interventions: Drug: Sodium Ozagrel

INTERVENTIONS:
Drug: Edaravone — Edaravone, at 30 mg, is intravenously administered by drip over 30 minutes b.i.d., in the morning and the evening.
  Other Names: Radicut
  Arms: Edaravone
Drug: Sodium Ozagrel — Sodium Ozagrel, at 80 mg, is intravenously administered by drip over 2 hours b.i.d., in the morning and the evening.
  Arms: Ozagrel

SUMMARY:
This study is randomized, Sodium Ozagrel (Thromboxane A2 Synthase Inhibitor) controlled study on acute ischemic stroke. The primary endpoints were the rate of patients with modified Rankin Scale score of 0-1 at 3 months.

ELIGIBILITY:
Inclusion Criteria:

1. Patients can be receive drug treatment within 24 hours after stroke onset
2. Patients with a level of consciousness between 0 (alert) and 3 (unable to recall name and date of birth) according to the Japan Coma Scale
3. Patients with motor dysfunction of upper and/or lower extremities
4. Patients aged 20 years or older when giving informed consent

Exclusion Criteria:

1. Serum creatinine of >1.5 mg/dL
2. Embolic infarction
3. Intracranial haemorrhage
4. Large infarction with severe consciousness
5. Transient ischemic attack (TIA)
6. A modified Rankin Scale score of ≥2 before stroke onset
7. Patients were receive drug treatment (argatroban, urokinase, tissue plasminogen activator, heparin, warfarin sodium, aspirin, ticlopidine hydrochloride, cilostazol, edaravone and sodium ozagrel) after stroke onset
8. Patients were receive surgical treatment or intravascular treatment
9. With severe complications (cirrhosis, heart failure, etc.)
10. Treating malignant tumor
11. Pregnant or possibly pregnant women, nursing mothers
12. History of edaravone, sodium ozagrel and ozagrel hydrochloride sensitivity
13. Less than 3 months since any other clinical trial or postmarketing study

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 401 (Actual)
Dates: Start 2004-08; Study Completion 2006-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yukito Shinohara, MD, Study Chair — Federation of National Public Service Personnel Mutual Aid Associations Tachikawa Hospital

REFERENCES:
- [Result] Shinohara Y, Saito I, Kobayashi S, Uchiyama S. Edaravone (radical scavenger) versus sodium ozagrel (antiplatelet agent) in acute noncardioembolic ischemic stroke (EDO trial). Cerebrovasc Dis. 2009;27(5):485-92. doi: 10.1159/000210190. Epub 2009 Mar 26. PMID 19321945

RESULTS

PARTICIPANT FLOW:
Groups:
- Ozagrel: Sodium Ozagrel, at 80 mg, is intravenously administered by drip over 2 hours b.i.d., in the morning and the evening.
Period: Overall Study
Arm/Group | Edaravone | Ozagrel
Started | 199 | 202
Safety Analysis Set | 194 | 198
Completed | 191 | 195
Not Completed | 8 | 7
Not completed — Lack of Efficacy | 3 | 3
Not completed — Protocol Violation | 4 | 4
Not completed — Nontreatment | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Edaravone | Ozagrel | Total
Number analyzed (Participants) | 191 | 195 | 386
Age, Customized [Number; unit: years]
  birth-19 years | 0 | 0 | 0
  20-64 years | 64 | 58 | 122
  65- years | 127 | 137 | 264
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 70 | 77 | 147
  Male | 121 | 118 | 239

OUTCOME MEASURES:

1. Secondary Outcome: Barthel Index Score
Description: The Barthel Index of Activities of Daily Living measures functional disability by quantifying patient performance in 10 activities of daily life. These activities can be grouped according to self-care (feeding, grooming, bathing, dressing, bowel and bladder care, and toilet use) and mobility (ambulation, transfers, and stair climbing). 5-point increments are used in scoring, with a maximal score of 100 indicating that a patient is fully independent in physical functioning, and a lowest score of 0 representing a totally dependent bed-ridden state.
  The number of patients with 95-100 Barthel Index was evaluated at at 3 months after treatment initiation.
Time Frame: 3 months
Measure: Number; unit: participants
Arm/Group | Edaravone | Ozagrel
Number analyzed (Participants) | 191 | 195
participants | 148 | 133

2. Secondary Outcome: Baseline NIH Stroke Scale Score
Description: The NIH stroke scale is a systematic assessment tool that provides a quantitative measure of stroke-related neurologic deficit. Values range from 0 (no deficit) to 42(dead).
Time Frame: Before treatment initiation
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Edaravone | Ozagrel
Number analyzed (Participants) | 191 | 195
scores on a scale | 3.7 (2.3) | 3.8 (2.7)

3. Secondary Outcome: NIH Stroke Scale Score at 14 Days
Description: The NIH stroke scale is a systematic assessment tool that provides a quantitative measure of stroke-related neurologic deficit. Values range from 0 (no deficit) to 42(dead). The number of patients with NIH stroke scale score of 0-1 at 14 days after treatment initiation.
Time Frame: 14 days
Measure: Number; unit: participants
Arm/Group | Edaravone | Ozagrel
Number analyzed (Participants) | 190 | 193
participants | 98 | 108

4. Secondary Outcome: NIH Stroke Scale Score at 1 Month
Description: The NIH stroke scale is a systematic assessment tool that provides a quantitative measure of stroke-related neurologic deficit. Values range from 0 (no deficit) to 42(dead). The number of patients with NIH stroke scale score of 0-1 at 1 month after treatment initiation.
Time Frame: 1 month
Measure: Number; unit: participants
Arm/Group | Edaravone | Ozagrel
Number analyzed (Participants) | 190 | 195
participants | 117 | 119

5. Primary Outcome: the Rate of Patients With a Modified Rankin Scale Score of 0-1
Description: The number of patients with mRS score of 0-1 (good outcome) at 3 months after treatment initiation. The mRS has 6 items, where 0 = No symptoms at all, 1 = No significant disability despite symptoms, 2 = Slight disability, 3 = Moderate disability, 4 = Moderately severe disability, 5 = Severe disability. The higher scores reflect increased disability.
Time Frame: 3 months
Measure: Number; unit: participants
Arm/Group | Edaravone | Ozagrel
Number analyzed (Participants) | 191 | 195
participants
  Score(0-1) | 109 | 98
  0 | 46 | 39
  1 | 63 | 59
  2 | 37 | 40
  3 | 22 | 29
  4 | 19 | 24
  5 | 2 | 3
  Death | 2 | 1

6. Secondary Outcome: NIH Stroke Scale Score at 3 Months
Description: The NIH stroke scale is a systematic assessment tool that provides a quantitative measure of stroke-related neurologic deficit. Values range from 0 (no deficit) to 42(dead). The number of patients with NIH stroke scale score of 0-1 at 3 months after treatment initiation.
Time Frame: 3 months
Measure: Number; unit: participants
Arm/Group | Edaravone | Ozagrel
Number analyzed (Participants) | 191 | 195
participants | 135 | 140

7. Secondary Outcome: Japan Stroke Scale (Motor Function) Score at 14 Days
Description: The Japan stroke scale (motor function) is a systematic assessment tool that provides a quantitative measure of stroke-related neurologic deficit. Values range from -0.26 (no deficit) to 31.29 (worst). The mean of Japan stroke scale (motor function) score at 14 days after treatment initiation.
Time Frame: 14 days
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Edaravone | Ozagrel
Number analyzed (Participants) | 190 | 193
units on a scale | 4.521 (6.651) | 4.686 (6.872)

8. Secondary Outcome: Japan Stroke Scale (Motor Function) Score at 1 Month
Description: The Japan stroke scale (motor function) is a systematic assessment tool that provides a quantitative measure of stroke-related neurologic deficit. Values range from -0.26 (no deficit) to 31.29 (worst). The mean of Japan stroke scale (motor function) score at 1 month after treatment initiation.
Time Frame: 1 month
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Edaravone | Ozagrel
Number analyzed (Participants) | 190 | 195
units on a scale | 3.632 (6.086) | 3.680 (5.885)

9. Secondary Outcome: Japan Stroke Scale (Motor Function) Score at 3 Months
Description: The Japan stroke scale (motor function) is a systematic assessment tool that provides a quantitative measure of stroke-related neurologic deficit. Values range from -0.26 (no deficit) to 31.29 (worst). The mean of Japan stroke scale (motor function) score at 3 months after treatment initiation.
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Edaravone | Ozagrel
Number analyzed (Participants) | 189 | 194
units on a scale | 2.507 (5.232) | 2.927 (5.361)

10. Secondary Outcome: Modified Rankin Scale Score
Description: The number of patients with an Modified Rankin Scale score of 0-1 was evaluated at 6 months after treatment initiation. The Modified Rankin Scale has 6 items, where 0 = No symptoms at all, 1 = No significant disability despite symptoms, 2 = Slight disability, 3 = Moderate disability, 4 = Moderately severe disability, 5 = Severe disability. The higher scores reflect increased disability.
Time Frame: 6 months
Measure: Number; unit: participants
Arm/Group | Edaravone | Ozagrel
Number analyzed (Participants) | 186 | 193
participants | 112 | 108

ADVERSE EVENTS:
Arm/Group | Edaravone | Ozagrel
Serious Adverse Events (participants affected / at risk) | 27/194 | 28/198
Other Adverse Events (participants affected / at risk) | 102/194 | 107/198
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Edaravone (N=194) | Ozagrel (N=198)
Anastomotic ulcer haemorrhage (Injury, poisoning and procedural complications) | 1 | 0
Angina pectoris (Cardiac disorders) | 1 | 0
Anti-neutrophil cytoplasmic antibody positive vasculitis (Immune system disorders) | 1 | 0
Arrhythmia (Cardiac disorders) | 1 | 0
Arteriosclerosis (Vascular disorders) | 0 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Brain herniation (Injury, poisoning and procedural complications) | 0 | 1
Cardiac failure (Cardiac disorders) | 0 | 1
Carpal tunnel syndrome (Nervous system disorders) | 0 | 1
Cerebral haemorrhage (Nervous system disorders) | 1 | 0
Cerebral infarction (Nervous system disorders) | 5 | 11
Constipation (Gastrointestinal disorders) | 0 | 1
Depression (Psychiatric disorders) | 1 | 0
Duodenal ulcer (Gastrointestinal disorders) | 1 | 0
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 1 | 0
Erysipelas (Infections and infestations) | 0 | 1
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 | 0
Femur fracture (Injury, poisoning and procedural complications) | 1 | 0
Haemorrhagic cerebral infarction (Nervous system disorders) | 0 | 1
Hemiplegia (Nervous system disorders) | 0 | 2
Ileus (Gastrointestinal disorders) | 2 | 0
Inguinal hernia (Gastrointestinal disorders) | 1 | 0
Liver disorder (Hepatobiliary disorders) | 0 | 1
Loss of consciousness (Nervous system disorders) | 0 | 1
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Pelvic fracture (Injury, poisoning and procedural complications) | 1 | 0
Pharyngitis (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 2 | 1
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Psychotic disorder due to a general medical condition (Psychiatric disorders) | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Renal failure acute (Renal and urinary disorders) | 0 | 1
Sciatica (Nervous system disorders) | 0 | 1
Shock haemorrhagic (Vascular disorders) | 0 | 1
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 | 1
Thrombotic stroke (Nervous system disorders) | 1 | 0
Transient ischemic attack (Nervous system disorders) | 2 | 0
Upper limb fracture (Injury, poisoning and procedural complications) | 0 | 1
Urinary tract infection (Infections and infestations) | 1 | 1
Vertigo (Ear and labyrinth disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Edaravone (N=194) | Ozagrel (N=198)
Constipation (Gastrointestinal disorders) | 59 | 64
Diarrhea (Gastrointestinal disorders) | 10 | 6
Headache (Nervous system disorders) | 11 | 12
Insomnia (Psychiatric disorders) | 24 | 33
Nasopharyngitis (Infections and infestations) | 19 | 13
Pruritus (Skin and subcutaneous tissue disorders) | 9 | 10
Urinary tract infection (Infections and infestations) | 9 | 11
Back pain (Musculoskeletal and connective tissue disorders) | 11 | 17

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other